CLINICAL TRIAL: NCT05732857
Title: Perioperative Effects of Valveless Trocar Versus Standard Trocar in Robot-assisted Complex Partial Nephrectomy: a Randomized Prospective Study
Brief Title: Valveless Trocar Versus Standard Trocar in Robot-assisted Complex Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, MD, E Forastiere, MD, Head of Anestesiology and Intensive care Unit, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1795/22
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cancer of Kidney
Keywords: robotic nephrectomy; pneumoperitoneum; trocar valveless; general anesthesia; mechanical ventilation
MeSH Terms: conditions — Kidney Neoplasms; Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: control arm: patients in which traditional laparoscopic trocar is used intervention arm: patients in which the valveless trocar is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trocar standard (Sham Comparator): patients in whom the standard trocar will be used to perform robot-assisted complex partial nephrectomy surgery
  Interventions: Device: standard trocar
- trocar valveless (Active Comparator): patients in whom the valveless trocar will be used to perform robot-assisted complex partial nephrectomy surgery
  Interventions: Device: valveless trocar

INTERVENTIONS:
Device: valveless trocar — the valveless trocar will be used instead of the standard trocar - these trocars are used for insufflation of carbon dioxide into the abdomen
  Other Names: airseal
  Arms: trocar valveless
Device: standard trocar — standard trocar, usually camera port for robotic surgery
  Arms: trocar standard

SUMMARY:
The goal of this clinical trial is to compare two kind of trocar in patients undergoing complex robot-assisted partial nephrectomy. The main question it intends to answer is whether the use of valveless trocars can significantly reduce carbon dioxide absorption.

DETAILED DESCRIPTION:
In the literature there are studies on the benefit of valveless trocars in robotic surgery. There are no studies on the potential effects even in complex kidney surgery. Through this randomized study we want to investigate whether the ability to clear CO2 is better using valveless trocars

ELIGIBILITY:
Inclusion Criteria:

* asa status 1-3
* surgical classification RENAL or PADUA score >9

Exclusion Criteria:

* BMI>30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
carbon dioxide elimination rate: using the formula where end tidal carbon dioxide multiplied by minute volume divided by arterial pressurea (760mmHg) multiplied by patient weight | before extubation

SECONDARY OUTCOMES:
postoperative acute pain: using the NRS scale | at 1 hour and at 4 hour after the end of surgery
subcutaneous emphysema: through clinical observation at the end of the intervention | at 30 minutes afetr the end of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, IRCCS Regina Elena National Cancer Institute, Roma, Italy